CLINICAL TRIAL: NCT04942327
Title: How Well Informed is a Otorhynolaryngologist in a Secondary Setting About the Hearing Enhancement Interventions and Reimbursement Criteria Related to Hearing Implants?
Brief Title: Awareness Among Hearing Enhancement Interventions and Reimbursement Criteria of Hearing Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Awareness
Record Dates: First submitted 2021-05-28; First posted 2021-06-28 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-05

CONDITIONS: Awareness; Hearing Impairment; Otorhinolaryngologic Surgical Procedures; Implant
MeSH Terms: conditions — Hearing Loss | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview (Other): This will be evaluated through a specific questionnaire that will be systematically gone over with the participants during an interview in the first and third phases.
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — This will be evaluated through a specific questionnaire that will be systematically gone over with the participants during an interview in the first and third phases.

SUMMARY:
The following research questions will be investigated:

What is the knowledge of medical interventions for moderate to severe hearing loss and what is the knowledge of the reimbursement criteria for hearing implants of otorhinolaryngologists in a secondary setting in Brabant. This will be evaluated by means of a specific questionnaire that will be systematically gone over with the participants during an interview in the first and third phase.

In a second phase, the investigators will investigate how the knowledge of medical interventions for moderate to severe hearing loss and the knowledge of the reimbursement criteria for hearing implants of otorhinolaryngologists in a secondary setting in Brabant can be increased by training the otorhinolaryngologists in a secondary setting in Brabant.

In the third phase, the investigators will evaluate the knowledge of hearing implant interventions and reimbursement criteria among otorhinolaryngologists in a secondary setting.

DETAILED DESCRIPTION:
In most developed economies, cochlear implants have been shown to be the most successful neuroprostheses for sensory moderate or severe neurosensory loss. These neuroprostheses are cost-effective with low complication rates. However, the literature indicates that there is a low level of awareness of the benefits of cochlear implants among the general population and among healthcare professionals. In addition, a lack of specific referral pathways has been reported. Utilization rates for adult hearing aids in people with severe or profound loss are 70% to 90%, but uptake in adults for cochlear implants is less than 10%.

Therefore, the aim of this research project is to investigate the knowledge about medical interventions in moderate to severe hearing loss and the knowledge about reimbursement criteria of hearing implants of otorhinolaryngologists in a secondary setting in Brabant.

The study group will consist of a maximum of 100 geographically selected otorhinolaryngologists aged 25-70 years in a secondary setting in Brabant. A subselection will be made from the reachable otorhinolaryngologists in the region of Brabant. Recruitment will be discontinued when a maximum of 100 otorhinolaryngologists has been reached. A specific questionnaire will be systematically reviewed with the participants during an interview in the first and third phase. There is no financial compensation for the participants.

ELIGIBILITY:
Inclusion Criteria:

* Otorhinolaryngologists working in a secondary setting
* Dutch and French speaking

Exclusion Criteria:

* Otorhinolaryngologists working in a tertiary setting attached to a university

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Behavior change: Questionnaire | through study completion, an average of 1 year
  Change in referral pattern
Knowledge: Questionnaire: | through study completion, an average of 1 year
  Increased knowledge of hearing implant interventions and reimbursement criteria among otorhinolaryngologists in a secondary setting.

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Topsakal, Professor, Principal Investigator — UZ Brussel / VUB
Locations (1):
- UZ Brussel, Brussels, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchman CA, Gifford RH, Haynes DS, Lenarz T, O'Donoghue G, Adunka O, Biever A, Briggs RJ, Carlson ML, Dai P, Driscoll CL, Francis HW, Gantz BJ, Gurgel RK, Hansen MR, Holcomb M, Karltorp E, Kirtane M, Larky J, Mylanus EAM, Roland JT Jr, Saeed SR, Skarzynski H, Skarzynski PH, Syms M, Teagle H, Van de Heyning PH, Vincent C, Wu H, Yamasoba T, Zwolan T. Unilateral Cochlear Implants for Severe, Profound, or Moderate Sloping to Profound Bilateral Sensorineural Hearing Loss: A Systematic Review and Consensus Statements. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):942-953. doi: 10.1001/jamaoto.2020.0998. PMID 32857157
- [Background] D'Haese PSC, De Bodt M, Van Rompaey V, Van de Heyning P. Awareness of Hearing Loss in Older Adults: Results of a Survey Conducted in 500 Subjects Across 5 European Countries as a Basis for an Online Awareness Campaign. Inquiry. 2018 Jan-Dec;55:46958018759421. doi: 10.1177/0046958018759421. PMID 29529899
- [Background] Sorkin DL. Access to cochlear implantation. Cochlear Implants Int. 2013 Mar;14 Suppl 1(Suppl 1):S1. doi: 10.1179/1467010013Z.00000000081. No abstract available. PMID 23453144
- See also: Background information — http://www.researchgate.net/publication/333894238_The_Need_to_Increase_Awareness_and_Access_to_Cochlear_Implantation